CLINICAL TRIAL: NCT05483465
Title: Effects of NAD Restoration on Neurovascular Coupling in Community Dwelling Older Adults
Brief Title: The Effect of NAD Supplementation on Brain Vascular Health in Aging
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: University of Pennsylvania (Other); Oklahoma Medical Research Foundation (Other); Elysium Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14782
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Aging
Keywords: NAD; NR; nicotinamide riboside; neurovascular coupling; endothelial function; cognitive function
MeSH Terms: interventions — nicotinamide-beta-riboside; Sugars

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, parallel study design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All data will be unmasked upon completion of the trial, or during performance of data review if requested by the data safety and monitoring board.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NR (Experimental): Treatment with oral NR (1g/day per os for 8 weeks)
  Interventions: Drug: Nicotinamide riboside
- Control (Placebo Comparator): Visually identical placebo (daily, per os, for 8 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide riboside — Oral NR, 1g/day per os for 8 weeks
  Other Names: NR
  Arms: NR
Drug: Placebo — Visually identical pill to NR, daily per os for 8 weeks
  Other Names: Sugar pill
  Arms: Control

SUMMARY:
Daily consumption of one of the forms of Vitamin B3, the Nicotinamide Riboside (NR), energizes the body and combats cellular aging. This study is designed to test whether NR can also improve brain health and memory.

DETAILED DESCRIPTION:
This study is designed to test the hypothesis that restoration of Nicotinamide Adenine Dinucleotide (NAD) levels with Nicotinamide Riboside (NR) in older adults will improve neurovascular coupling (NVC) responses and micro- and macrovascular endothelial function. This hypothesis will be tested by assessing the effects of treatment with oral NR (1g/day per os for 8 weeks) or placebo (8 weeks) in community dwelling older adults (60-85 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 and ≤85 years of age
* Adequate hearing and visual acuity to participate in the examinations
* Ability to read and write in English
* Competence to provide informed consent.
* Mini-Mental State Exam score ≥24

Exclusion Criteria:

* Vision or hearing impairment that would impair the ability to complete study assessments
* Active CNS disease including multiple sclerosis, uncontrolled seizures, active brain cancer
* Cerebrovascular accident other than TIA within 60 days prior to Visit 0
* Major psychiatric disease, including major depression not currently controlled on medications, alcohol or drug abuse
* Abnormal kidney function (creatinine >2mg/dL or EGFR <30mL/min) by most recent labs within 6 months prior to Visit 0
* Elevated liver enzymes (AST and/or ALT above x2 upper limit of normal) by most recent labs within 6 months prior to Visit 0
* Treatment with other NAD enhancers (Nicotinamide riboside or nicotinamide mononucleotide) within 4 weeks prior to randomization.
* Any other medical condition which, in the opinion of investigator, would render the patient inappropriate or too unstable to complete the study protocol

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in neurovascular coupling using functional near infrared spectroscopy (fNIRS) | 8 weeks
  Functional near infrared spectroscopy (fNIRS) will be performed during the cognitive n-back task. fNIRS approach generates data that represent a relative change in oxygenated and deoxygenated hemoglobin measured over the cortical brain tissues. Neurovascular coupling will be evaluated as a change in oxy- and deoxy-hemoglobin between before and after treatment. Units of measure - beta. Reported as a %change from baseline, before and after treatment.
Change in neurovascular coupling using transcranial Doppler | 8 weeks
  Transcranial Doppler sonography will be used to measure the change in the blood flow velocities during the cognitive n-back task between before and after treatment. Units of measure - % change between the n-back tasks. Reported as a %change from baseline, before and after treatment.
Change in neurovascular coupling using the dynamic retinal vessel analysis | 8 weeks
  Flicker light-induced dilation of the retinal vessels (percentage increase over baseline diameter) will be measured in the right or left eye of each study participant using the Dynamic Vessel Analyzer (DVA, IMEDOS Systems, Jena, Germany). Units of measure mm, reported as a %change from baseline, before and after treatment.
Change in neuronal activity | 8 weeks
  EEG signal will be collected to generate spectral data. These data will be used for comparison of EEG activity between before and after treatment. Units of measure - power spectral density. Reported as a %change from baseline, before and after treatment.

SECONDARY OUTCOMES:
Change in microvascular endothelial function | 8 weeks
  Changes in microvascular endothelial function will be assessed using laser speckle contrast imaging (LSCI) in the hand using the flow mediated dilation approach. The change in skin perfusion is calculated and reported as a %change from baseline, between before and after treatment. Units of measure - perfusion index (arbitrary units). Reported as a %change from baseline, before and after treatment.
Change in macrovascular endothelial function | 8 weeks
  Changes in macrovascular endothelial function will be assessed using sonography during flow mediated dilation approach. The change in brachial artery diameter (mm) is calculated and reported as a %change from baseline, between before and after treatment.
Change in deep tissue oxygen saturation | 8 weeks
  Transcutaneous deep tissue oxygen saturation will be measured using the inSpectra near infrared device. The data are calculated and reported as a %change from baseline, between before and after treatment.
Change in arterial stiffness | 8 weeks
  The arterial stiffness will be measured using the pulse wave analysis approach (SphygmoCor, Atcor medical, Itasca IL, or similar). Analysis generates the augmentation index which will be used for comparison before and after treatment.
Change in ECG | 8 weeks
  ECG will be recorded for heart rate variability analysis. The values of high frequency domain, low frequency domain, their ratio, as well as total power will be calculated and used for comparison before and after treatment.
Change in Glycocalyx - perfused boundary region | 8 weeks
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include perfused boundary region (um), and will be used for comparison before and after treatment.
Change in capillary density | 8 weeks
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include capillary density (mm/mm^2), and will be used for comparison before and after treatment.
Change in red blood cell velocity | 8 weeks
  Video recordings of the sublingual vasculature will be performed using the high definition video camera GlycoCheck (Microvascular health solutions). Data collected will include red blood cell velocity (um/sec), and will be used for comparison before and after treatment.
Change in Attention | 8 weeks
  The allocation of one's limited capacities to deal with an abundance of environmental stimulation will be measured in a combined "Flanker Inhibitory Control and Attention Test".Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Episodic Memory | 8 weeks
  Cognitive processes involved in the acquisition, storage and retrieval of new information, will be measured using the "Picture Sequence Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Working Memory | 8 weeks
  The ability to store information until the amount of information to be stored exceeds one's capacity to hold that information will be measured using the "List Sorting Working Memory Test". Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Language | 8 weeks
  Picture Vocabulary Test measures receptive vocabulary administered in a computer-adaptive test (CAT) format. Respondents select the picture that most closely matches the meaning of the word, before and after treatment. Unit of measure - overall score (bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Executive Function | 8 weeks
  The capacity to plan, organize and monitor the executive of behaviors that are strategically directed in a goal-oriented manner will be measured using the "Dimensional Change Card Sort Test". Units of measure - score (from 0 to 10, bigger number is better). Reported as a %change from baseline, before and after treatment.
Change in Processing Speed | 8 weeks
  Pattern Comparison Processing Speed Test assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed. Units of measure - score (from 0 to 130, bigger number is better). Reported as a %change from baseline, before and after treatment.
Blood collection | 8 weeks
  Blood samples will be collected to measure concentration of NAD metabolites for comparison before and after treatment. Blood samples will also be used in in vitro assays to measure the effect of treatment on endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Andriy Yabluchanskiy, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
The results may be uploaded to scientific online repositories such as PhysioNet (or other) as requested by the journal when data is submitted for publication. In that case, all data will be de-identified and labeled by group+number (for example Placebo1, Placebo2, NR1, NR2, these IDs will be different from study IDs stored on the servers at the OUHSC) and supported by subjects' age, sex, comorbidities and treatments data.